CLINICAL TRIAL: NCT00777894
Title: External Beam Radiotherapy for Unresectable Hepatocellular Carcinoma. A Multicenter Phase I/II Trial.
Brief Title: Radiation Therapy in Treating Patients With Liver Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 77/07; SWS-SAKK-77/07; EU-20884; SWS-SASL-26
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Liver Cancer
Keywords: advanced adult primary liver cancer; localized unresectable adult primary liver cancer; adult primary hepatocellular carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiation: 3-dimensional conformal radiation therapy (Experimental)
  Interventions: Radiation: 3-dimensional conformal radiation therapy; Radiation: intensity-modulated radiation therapy; Radiation: stereotactic body radiation therapy

INTERVENTIONS:
Radiation: 3-dimensional conformal radiation therapy — Once daily RT sessions with 2 Gy, five days a week (on weekdays), will be performed.
  Phase I: Dose finding according to the following escalation table:
  Dose level Radiotherapy dose (1 x 2 Gy session/day, 5 sessions/week)
  1. (3 patients) 27 x 2 Gy = 54 Gy
  2. (3 patients) 29 x 2 Gy = 58 Gy, with optional field reduction after a dose of 54 Gy
  3. (3 patients) 31 x 2 Gy = 62 Gy, with optional field reduction after a dose of 54 Gy
  4. (5 patients) 33 x 2 Gy = 66 Gy, with optional field reduction after a dose of 54 Gy
  5. (5 patients) 35 x 2 Gy = 70 Gy, with optional field reduction after a dose of 54 Gy
  Phase II: The dose for phase II will be recommended according to the MTD determined in phase I, if the MTD is 62 Gy or higher. If the MTD is 58 Gy or lower, the phase II part of the trial will not be performed.
Radiation: intensity-modulated radiation therapy — Once daily RT sessions with 2 Gy, five days a week (on weekdays), will be performed.
  Phase I: Dose finding according to the following escalation table:
  Dose level Radiotherapy dose (1 x 2 Gy session/day, 5 sessions/week)
  1. (3 patients) 27 x 2 Gy = 54 Gy
  2. (3 patients) 29 x 2 Gy = 58 Gy, with optional field reduction after a dose of 54 Gy
  3. (3 patients) 31 x 2 Gy = 62 Gy, with optional field reduction after a dose of 54 Gy
  4. (5 patients) 33 x 2 Gy = 66 Gy, with optional field reduction after a dose of 54 Gy
  5. (5 patients) 35 x 2 Gy = 70 Gy, with optional field reduction after a dose of 54 Gy
  Phase II: The dose for phase II will be recommended according to the MTD determined in phase I, if the MTD is 62 Gy or higher. If the MTD is 58 Gy or lower, the phase II part of the trial will not be performed.
Radiation: stereotactic body radiation therapy — Once daily RT sessions with 2 Gy, five days a week (on weekdays), will be performed.
  Phase I: Dose finding according to the following escalation table:
  Dose level Radiotherapy dose (1 x 2 Gy session/day, 5 sessions/week)
  1. (3 patients) 27 x 2 Gy = 54 Gy
  2. (3 patients) 29 x 2 Gy = 58 Gy, with optional field reduction after a dose of 54 Gy
  3. (3 patients) 31 x 2 Gy = 62 Gy, with optional field reduction after a dose of 54 Gy
  4. (5 patients) 33 x 2 Gy = 66 Gy, with optional field reduction after a dose of 54 Gy
  5. (5 patients) 35 x 2 Gy = 70 Gy, with optional field reduction after a dose of 54 Gy
  Phase II: The dose for phase II will be recommended according to the MTD determined in phase I, if the MTD is 62 Gy or higher. If the MTD is 58 Gy or lower, the phase II part of the trial will not be performed.

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. This may be an effective treatment for liver cancer.

PURPOSE: This phase I/II trial is studying the side effects and best dose of external-beam radiation therapy in treating patients with liver cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the feasibility and safety of radiotherapy (RT) in patients with hepatocellular carcinoma. (Phase I)
* To assess the safety and efficacy of RT in these patients. (Phase II)
* To generate reproducible peptide patterns of the serum proteome or specific serum sub proteomes in these patients.
* To assess changes in the proteome or sub proteome patterns after RT in these patients.
* To detect peptides that discriminate between before and after RT in these patients.
* To identify these discriminating peptides in these patients.

OUTLINE: This is a multicenter, phase I dose-escalation study followed by a phase II study.

Patients undergo radiotherapy (RT) once daily, five days a week, for 6 weeks. Intensity-modulated, 3-dimensional conformal, or fractionated stereotactic RT may be used.

After completion of study therapy, patients in the phase I portion are followed for 1 year and patients in the phase II portion are followed for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically, cytologically, or radiologically confirmed hepatocellular carcinoma

  * Clinical stage T2-4, N0-1, M0 (stage II, IIIA, IIIB, IIIC) OR unresectable T1, N0-1, M0 (stage I) disease

    * M1 disease allowed in phase I if at least 90% of the tumor load (volume) is in the liver
* Measurable disease (at least one liver lesion that can be measured in at least one dimension as ≥ 10 mm in multislice CT scan/MRI)
* Volumetry of liver tumor and residual liver tissue: residual liver volume (= total liver volume - gross tumor volume) has to be ≥ 800 mL and ≥ 40% of total liver volume
* No operable disease (with curative intent or planned liver transplantation)
* No presence of clinical ascites

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Cirrhosis Child-Pugh class A or B (Child-Pugh score of ≤ 9)
* Hemoglobin ≥ 100 g/L
* ANC ≥ 1,200/mm³
* Platelet count ≥ 50,000/mm³
* ALT and AST ≤ 7 times upper limit of normal (ULN)
* AP ≤ 10 times ULN
* Bilirubin ≤ 50 μmol/L
* INR ≤ 2
* Creatinine clearance ≥ 50 mL/min
* Functional left kidney (scintigraphy mandatory for phase I, phase II only if indicated)
* Lipase ≤ 2 times ULN (phase I only)
* Able to tolerate proton-pump inhibitors or H2 antagonists during radiation therapy
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 months after completion of study therapy
* No prior malignancy allowed, except for the following:

  * Adequately treated cervical carcinoma in situ
  * Adequately treated localized nonmelanoma skin cancer
  * Any other malignancy from which patient has been disease-free for 5 years
* No presence of medically uncontrolled encephalopathy
* No myocardial infarction within the past 6 months
* No esophageal varices ≥ grade 3, with red signs, or bleeding within the past 3 months
* No symptoms of colitis, enteritis, esophagitis, fistula, gastritis, ileus, necrosis, perforation, stricture, or ulcer
* No severe anorexia, constipation, dehydration, diarrhea, or vomiting
* No serious underlying medical condition that, in the opinion in the investigator, would preclude study participation (e.g., active autoimmune disease or uncontrolled diabetes)

  * Portal vein thrombosis allowed
* No psychiatric disorder precluding understanding of information on study related topics or giving informed consent
* No nutritional intake < 1500 calories per day (corrected)
* No weight loss ≥ 15 % within the past 3 months

PRIOR CONCURRENT THERAPY:

* At least 8 weeks since prior transarterial chemoembolization (TACE), radiofrequency ablation, or radiotherapy (RT) unless progressive disease was documented after this therapy
* At least 21 days since prior and no other concurrent treatment with experimental drugs
* At least 21 days since prior and no other concurrent treatment on another clinical trial
* At least 21 days since prior and no other concurrent anticancer therapy
* No prior RT to the abdomen or caudal chest

  * Prior RT to pelvis allowed
  * Prior RT to chest must be above D5 vertebra
  * Portal vein embolization ligation or pre-RT TACE allowed
* No concurrent treatment with steroids or non-steroidal anti-inflammatory drugs during RT (proton-pump inhibitor allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-11; Primary Completion 2014-01 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (Phase I) | during RT or within 30 days after the last RT dose, is a DLT.
Best objective response of target liver lesions (TLLs) | according to RECIST criteria for up to 1 year after completion of study therapy (Phase II)

SECONDARY OUTCOMES:
Best objective response of TLLs according to RECIST criteria (Phase I) | according to RECIST criteria (Phase I)
Adverse events according to NCI CTCAE v.3.0 | during therapy and within 3 months after completion of study therapy (Phases I and II)
Volumetric response of TLLs | at 5 months after completion of study therapy (Phase II)
Time to progression of TLLs (Phase II) | calculated from registration until documented tumor progression of target liver lesions.
Duration of response of TLLs (Phase II) | the time from achieving an objective response (CR + PR) to a progression of target liver lesions according to RECIST or death.
Stable disease of TLLs (Phase II) | will be determined according to RECIST
Time to liver event (Phase II) | from registration until progressive liver disease.
Progression-free survival (Phase II) | calculated from registration until documented tumor progression or death, whichever occurs first.
Overall survival (Phase II) | calculated from registration until death
Compensatory liver tissue hypertrophy at baseline and at 5 months after completion of study therapy (Phase II) | Increase in residual liver volume (= total liver - GTV) (ml) between registration and 5 months after RT will be calculated
Child-Pugh Score | at last study visit and at 1, 2, 3, and 5 months after completion of study therapy (Phase II)
Serum alpha-fetoprotein level (Phase II) | will be measured until progression, if AFP is ≥ 1.5 x ULN at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Naehrig, MD, Study Chair — Unviersitaetsspital Basel; Ilja Frank Ciernik, MD, Study Chair — Städtisches Klinikum Dessau; Daniel Aebersold, MD, Study Chair — Insel Gruppe AG, University Hospital Bern; Jean-Francois Dufour, MD, Study Chair — Insel Gruppe AG, University Hospital Bern
Locations (6):
- Maastro Lab at University of Maastricht, Maastricht, Netherlands
- Switzerland (5):
  - Kantonsspital Aarau, Aarau
  - Universitaetsspital-Basel, Basel
  - Istituto Oncologico della Svizzera Italiana - Ospedale San Giovanni, Bellinzona
  - Inselspital Bern, Bern
  - Kantonsspital - St. Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Herrmann E, Naehrig D, Sassowsky M, Bigler M, Buijsen J, Ciernik I, Zwahlen D, Pellanda AF, Meister A, Brauchli P, Berardi S, Kuettel E, Dufour JF, Aebersold DM; Swiss Group for Clinical Cancer Research (SAKK). External beam radiotherapy for unresectable hepatocellular carcinoma, an international multicenter phase I trial, SAKK 77/07 and SASL 26. Radiat Oncol. 2017 Jan 13;12(1):12. doi: 10.1186/s13014-016-0745-0. PMID 28086942